CLINICAL TRIAL: NCT02154867
Title: Recalibrating Intestinal Microflora in IBS by Fecal Transplantation
Brief Title: Fecal Microbial Transplantation in Treatment of Irritable Bowel Syndrome; a Double Blinded Placebo Controlled Trial.
Acronym: REFIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013/971/REK
Record Dates: First submitted 2014-04-10; First posted 2014-06-03 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS-D; FMT; metagenomics; gut microbiome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fecal transplantation (Experimental): Fecal transplantation of freshly prepared feces from healthy donor. Application by colonoscope in proximal half of colon.
  Interventions: Biological: Fecal transplantation
- Placebo fecal transplantation (Placebo Comparator): Sham transplant subject's own feces. Application by colonoscope in proximal part of colon.
  Interventions: Other: Placebo fecal transplant

INTERVENTIONS:
Biological: Fecal transplantation — Preparation of flesh feces by blending in 0.9 % saline and crude filtering. The solution is applied in proximal colon of IBS patient by colonoscopy after standard bowel preparation.
  Other Names: Fecal microbial transplantation
  Arms: Fecal transplantation
Other: Placebo fecal transplant — Fecal transplantation with own feces
  Arms: Placebo fecal transplantation

SUMMARY:
Fecal Microbial Transplantation in Treatment of Irritable Bowel Syndrome; a Double Blinded Placebo Controlled Trial - the REFIT project

Irritable bowel syndrome (IBS) is a condition characterized by variable complaints like diarrhoea, bloating and abdominal pain, and may result in considerably reduced quality of life and increased sickness absence. The prevalence of IBS in the general population may be as high as 15 per cent depending on the diagnostic criteria used. The pathophysiology of IBS is poorly understood and theories of visceral hypersensitivity, micro-inflammation and other less well founded theories have been stated. So far, no measurement or test can affirm diagnosis, but exclusion of organic diseases in combination with a typical symptom pattern according to the Rome classification can set the diagnosis.

Earlier non-controlled case reports have shown a convincing effect of fecal microbial transplantation (FMT) in IBS patients. However, no placebo controlled trial has been performed in this condition. Changes in the gut microbiome may be an important factor in IBS pathogenesis. Microbiome analysis has revealed changes in microbiome composition that may trigger changes in visceral sensibility and pain perception.

The fecal microbial transplantation (FMT) procedure has been used primarily to treat clostridium difficile infections. Few minor side effects have been reported.

Hypothesis: IBS is caused by an imbalance of the gut microbiome that may be reset by transplanting a microbiome sample from a healthy donor.

Aim of study:

* To test the clinical effect of FMT in patients with IBS
* To describe the fecal microbiome in IBS patients
* To describe changes in the fecal microbiome of IBS patients following FMT

The REFIT study will perform a randomized placebo-controlled double blinded trial of FMT on IBS according to the Rome 3 criteria. A study group of 60 IBS (diarrhoea variant) patients will recruited from general practice and allocated to active (30) or placebo (30) by block randomization. Donors will be 15 healthy volunteers with no risk behaviour and a pre-screening for communicable diseases will be performed.

Outcome measures will be clinical assessment by IBS-severity scoring system (IBS-SSS) at 0, 1, 3, 6, and 12 months. Microbiome analysis will be performed by metagenomic sequencing (University of Tromsø) at 0, 3, and 12 months for patients, and at inclusion for donors.

ELIGIBILITY:
Inclusion Criteria for patients:

* Patients with IBS-D according to Roma 3 criteria

Exclusion Criteria for patients:

* Immunomodulating medication
* Nocturnal abdominal pain
* Constant abdominal pain
* Alarm symptoms like rectal bleeding, weight loss, nightsweats
* Symptomatic heart/vascular/lung disease
* Renal failure
* Known food allergy
* Microscopic/collagenous colitis
* non-compliant
* BMI <18

Inclusion criteria for donors:

* healthy volunteers

Exclusion criteria for donors

* Tattoos, imprisoning or piercing last 3 months
* Any history of chronic diarrhoea, constipation, inflammatory bowel disease, irritable bowel disease, colorectal polyps or cancer, immunosuppression, morbid obesity, metabolic syndrome, atopica, or fatigue
* positive test for hepatitis B, C, HIV, treponema pallidum
* sexual high risk habits
* antibiotic treatment in the past 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-12; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in subjective symptom score | at 0 and 3 months
  Comparison of Irritable bowel syndrome severity scoring system (IBS-SSS) grade assessment before and after fecal transplantation

SECONDARY OUTCOMES:
Microbiome profile change | at 0, 3 and 12 months
  Characterization of fecal microbiome by metagenomic analysis before and after intervention
Long term effects of fecal transplantation | at 12 months
  Assessment of symptom burden by IBS-SSS
Safety of fecal transplantation in IBS | during study period (0-12 months)
  Registration of any adverse events. If any serious adverse events are encountered, the study group and local ethics committee will evaluate if study should be terminated.

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Goll, PhD, Principal Investigator — University Hospital of North Norway; Per C Valle, PhD, Study Director — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Harstad, Norway

REFERENCES:
- [Derived] Goll R, Johnsen PH, Hjerde E, Diab J, Valle PC, Hilpusch F, Cavanagh JP. Effects of fecal microbiota transplantation in subjects with irritable bowel syndrome are mirrored by changes in gut microbiome. Gut Microbes. 2020 Nov 9;12(1):1794263. doi: 10.1080/19490976.2020.1794263. PMID 32991818
- [Derived] Johnsen PH, Hilpusch F, Cavanagh JP, Leikanger IS, Kolstad C, Valle PC, Goll R. Faecal microbiota transplantation versus placebo for moderate-to-severe irritable bowel syndrome: a double-blind, randomised, placebo-controlled, parallel-group, single-centre trial. Lancet Gastroenterol Hepatol. 2018 Jan;3(1):17-24. doi: 10.1016/S2468-1253(17)30338-2. Epub 2017 Nov 1. PMID 29100842